CLINICAL TRIAL: NCT04671797
Title: Dinner Time 2: Effect of Delayed Eating or Sleeping on Metabolism
Acronym: DT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Arkansas (Other); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00156120-2
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: healthy volunteers; fat oxidation; sleep; circadian; glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Dinner first (Experimental): Participants will be served dinner and a stable isotope of palmitate to measure fat oxidation, at an early dinner time (DLMO-3h) followed by a sleep study (DLMO+2h). This arm will cross-over to the other 2 arms in random order.
  Interventions: Behavioral: Early dinner; Behavioral: Late Dinner; Behavioral: Late Dinner + Late Sleep
- Late Dinner first (Experimental): Participants will be served dinner and a stable isotope of palmitate to measure fat oxidation, at a late dinner time (DLMO+1h) followed by a sleep study (DLMO+2h). This arm will cross-over to the other 2 arms in random order.
  Interventions: Behavioral: Early dinner; Behavioral: Late Dinner; Behavioral: Late Dinner + Late Sleep
- Late Dinner + Late Sleep first (Experimental): Participants will be served dinner and a stable isotope of palmitate to measure fat oxidation, at a late dinner time (DLMO+1h) followed by delayed bedtime (DLMO+6h). This arm will cross-over to the other 2 arms in random order.
  Interventions: Behavioral: Early dinner; Behavioral: Late Dinner; Behavioral: Late Dinner + Late Sleep

INTERVENTIONS:
Behavioral: Early dinner — Dinner at DLMO-3, sleep at DLMO+2
Behavioral: Late Dinner — Dinner at DLMO+1, sleep at DLMO+2
Behavioral: Late Dinner + Late Sleep — Dinner at DLMO+1, sleep at DLMO+6

SUMMARY:
This study examines the acute impact of eating an "early" versus "late" dinner. "Early" and "late" will be customized to individuals based on the individuals' own circadian rhythms. Healthy adults will have the adults' circadian rhythm assessed by measuring the adults' dim light melatonin onset (DLMO). Based on the timing of DLMO, participants will be randomized to eating dinner before DLMO or after DLMO. The investigators will also compare the effects of delaying sleep relative to dinner time. Participants will eat meals in the laboratory and have serial plasma samples collected to examine profiles of free fatty acids, glucose, insulin, triglycerides, and oxidation of dietary fat.

DETAILED DESCRIPTION:
Obesity is a worldwide health problem. Recent studies suggest that the timing of meals may be critically important for weight control and cardiovascular health. Consuming calories later in the day is associated with greater risks of obesity, metabolic syndrome, and cardiovascular disease. Interventional diet studies also show more effective weight loss with early, rather than later eating. The investigators conducted a randomized crossover study comparing the metabolic effect of a "routine" dinner (RD,18:00) with that of an isocaloric "late" dinner (LD, 22:00) in 20 healthy volunteers. The investigators recently published results of this study, which the investigators now refer to as "Dinner Time 1". Relative to RD, LD increased post-dinner glucose peak by ~18% and lowered palmitate oxidation by ~10%. However, it is still unclear whether LD-induced impaired metabolic dysfunction is caused by eating at the "wrong" time relative to the body's central circadian clock, or it is caused by eating too close to bedtime, when sleep reduces metabolic demands.

To address this question, the investigators are now enlarging the scope of the present study, which the investigators now refer to as "Dinner Time 2". In Dinner Time 2, the investigators will examine the impacts of early dinner, late dinner, and the impact of delaying sleep after late dinner. The investigators will compare (1) the impact of early dinner time with later dinner time relative to DLMO with a routine sleep time; and (2) the impact of routine bedtime with late bedtime with a fixed late dinner time.

The investigators will examine the nocturnal and next-morning metabolic profile in a 3-arm randomized crossover study of healthy volunteers:

Arm 1: Early Dinner (dinner at DLMO-3, sleep at DLMO+2) Arm 2: Late Dinner (dinner at DLMO+1, sleep at DLMO+2) Arm 3: Late Dinner/Late Sleep (dinner at DLMO+1, sleep at DLMO+6)

The investigators will use serial blood sampling to assess the metabolic response to meals, and use an ingested stable isotope [(2H31)palmitate] tracer to calculate the oxidation of dietary lipid eaten at the different times.

ELIGIBILITY:
Inclusion:

* Healthy male and female adult volunteers, age 18-30
* BMI 18-30 kg/m2
* Accustomed to a bedtime before 1:00 A.M. or having mid-sleep on free days (MSF) earlier than 5 A.M. from the Munich Chronotype Questionnaire (MCTQ) (to exclude extreme late chronotypes)

Exclusions:

* Sleep disorder including insomnia, sleep apnea, circadian rhythm disorder, restless leg syndrome, narcolepsy, shift work sleep disorder
* Gastroesophageal reflux disease that affects ability to tolerate a dinner close to bed time.
* Chronic use of sedative hypnotics, anxiolytics, opiates
* Use of medications that can affect circadian rhythm (beta blockers, melatonin)
* Active smoking (may interfere with metabolism and Clinical Research Unit (CRU) activities)
* Diabetes (type 1 or 2)
* HbA1c point of care >= 6.5%
* Kidney disease
* Any known history of an inherited metabolic disorder
* Pregnant or lactating female (pregnancy test will be required)
* Professional or collegiate athlete
* Travel across >1 time zone within a 3-month period before and during the protocol
* DLMO > 24:00 will be excluded from the metabolic study visits

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Change in Glucose (mg/dl) | Baseline, 4 weeks and 8 weeks
  Serial blood samples taken during visit, 25 samples taken over 25 hours (One every hour) per visit.

SECONDARY OUTCOMES:
Change in Free Fatty Acids (FFA, mmol/L) | Baseline, 4 weeks and 8 weeks
  Serial blood samples taken during visit, 25 samples taken over 25 hours (One every hour) per visit.
Change in Insulin (mcU/ml) | Baseline, 4 weeks and 8 weeks
  Serial blood samples taken during visit, 25 samples taken over 25 hours (One every hour) per visit.
Change in Triglycerides (mg/dl) | Baseline, 4 weeks and 8 weeks
  Serial blood samples taken during visit, 25 samples taken over 25 hours (One every hour) per visit.
Change in Oxidation of palmitate (percent of isotope enrichment) | Baseline, 4 weeks and 8 weeks
  Serial blood samples taken during visit (14 samples per visit).
Change in melatonin [Dim light melatonin onset (DLMO)] | At 2 weeks prior to baseline (samples drawn every 30 minutes, up to 7 hours)
  Serial saliva samples taken during visit, 14 samples taken over 7 hours (one sample every 30 minutes) to access change in melatonin levels (pg/ml) over 7 hours.
Sleep architecture | Baseline, 4 weeks and 8 weeks
  Sleep stage distribution by EEG during each of the 3 sleep studies.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide raw data (without identifying information) to journals or other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be provided upon request within 1 year after publication and will be available to indefinitely.
Access Criteria: The PI will accept requests from other researchers who are examining pertinent outcomes.

REFERENCES:
- [Background] Gu C, Brereton N, Schweitzer A, Cotter M, Duan D, Borsheim E, Wolfe RR, Pham LV, Polotsky VY, Jun JC. Metabolic Effects of Late Dinner in Healthy Volunteers-A Randomized Crossover Clinical Trial. J Clin Endocrinol Metab. 2020 Aug 1;105(8):2789-802. doi: 10.1210/clinem/dgaa354. PMID 32525525
- See also: Study website — https://dinnertimestudy.net/